CLINICAL TRIAL: NCT01157715
Title: A Randomized, Double-masked, Multicenter, Controlled Dose- and Interval-ranging Clinical Study of Intravitreal Injection of KH902 in Patients With Neovascular Age-related Macular Degeneration (the AURORA Study)
Brief Title: A Randomized, Double-masked, Multicenter, Controlled Study of Intravitreal KH902 in Patients With Neovascular AMD
Acronym: AURORA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Collaborators: Beijing DMS Pharma Ltd. (Unknown); The Digital Angiography Reading Center (DARC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KHSWKH902001
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: KH902; age-related macular degeneration (AMD); choroidal neovascularization (CNV); intravitreal injection; best corrected visual acuity (BCVA); central retinal thickness
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 0.5 mg cohort (Experimental): patients will receive monthly intravitreal injections of 0.5 mg KH902 for 3 times in the study eye;following the initial 3-month fixed-dosing phase of the trial, patients will be randomized in a 1:1 ratio into one of two groups as follows: i. q1m group: patients will continue to receive monthly intravitreal injections of KH902 at the same dose received during the fixed dosing phase; ii. prn group: patients will continue to receive injection of KH902 at the same dose received during the fixed dosing phase, on an as needed (PRN) dosing schedule based upon the physician assessment of the need for re-treatment in accordance with pre-specified criteria .
  Interventions: Biological: intravitreal injection of KH902
- 2.0 mg cohort (Experimental): patients will receive monthly intravitreal injections of 2.0 mg KH902 for 3 times in the study eye;following the initial 3-month fixed-dosing phase of the trial, patients will be randomized in a 1:1 ratio into one of two groups as follows: i. q1m group: patients will continue to receive monthly intravitreal injections of KH902 at the same dose received during the fixed dosing phase; ii. prn group: patients will continue to receive injection of KH902 at the same dose received during the fixed dosing phase, on an as needed (PRN) dosing schedule based upon the physician assessment of the need for re-treatment in accordance with pre-specified criteria .
  Interventions: Biological: intravitreal injection of KH902

INTERVENTIONS:
Biological: intravitreal injection of KH902

SUMMARY:
This study is designed to access the safety and efficacy of multiple injections of KH902 at variable dosing regimens in patients with CNV due to neovascular AMD.

DETAILED DESCRIPTION:
AMD is the leading cause of severe vision loss in people over the age of 65 in the United States and other western countries. A quantity of documents indicate that neovascularization promoted by VEGF is main cause of visual acuity decline. Patients are starving for a new drug which can notably improve VA with less administration frequency and lower treatment cost.

The new drug Recombinant Human VEGF Receptor-Fc Fusion Protein (KH902) is a gene fusion protein. The pre-clinical researches and phase I study show that KH902 is effective and safe in inhibiting the growth, migration, pullulation of vascular endothelial cells and neovascularization induced by VEGF.

This study is designed to confirm the efficacy and safety of multiple injections of KH902 at variable dosing regimen in patients with CNV due to neovascular AMD. Based on the characteristics of KH902 and results from KH902 Phase I study as well as reference to clinical trials of similar drugs, it is determined that KH902 is administrated at 0.5mg/eye/time and 2.0mg/eye/time.

ELIGIBILITY:
Inclusion criteria:

* Signed the ICF; Age ≥ 50 years of either gender;
* Active primary or recurrent lesions with subfoveal or juxtafoveal CNV secondary to neovascular AMD in the study eye;
* Lesion size ≤ 12 disc areas in either eye;
* BCVA of the study eyes between 73 and 24 letters, inclusively, and the BCVA of fellow eyes ≥ 19 letters;
* Clear ocular media and adequate pupil dilation.
* If both eyes were eligible, only one was selected.

Exclusion criteria:

* History of vitreous hemorrhage, retinal detachment or macular hole, presence of retinal pigment epithelial tear, retinal macular traction or macular epiretinal membrane in the study eye;
* Subfoveal scar or atrophy in the study eye;
* Subretinal hemorrhage in the study eye;
* Uncontrolled glaucoma in either eye;
* Active inflammation or infection in either eye;
* Previous drug treatment, either anti-VEGF drugs or steroid derivatives, and/or, previous ophthalmologic operation or laser therapy in the study eye;
* History of surgery within one month preceding enrollment;
* Any uncontrolled clinical disorders;
* Patients of child-bearing potential do not adopted adequate contraception methods;
* Pregnant or nursing women;
* Patients need to exclude in the opinion of investigator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in BCVA | at 3-month
The incidence rate of adverse event | at 3-month

SECONDARY OUTCOMES:
Change from baseline in central retinal thickness | at 3-month and 12-month

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxin Li, MD, Prof., Principal Investigator — Peking University People's Hospital
Locations (9):
- China (9):
  - Optometry and Ophthalmology Hospital of Wenzhou Medical College, Wenzhou, Fujian
  - Zhongshan Ophthalmic Center, Sun-Yat University, Guangzhou, Guangdong
  - Second Affiliated Hospital of Xiangya Medical College, Changsha, Hunan
  - Xijing Hosiptal of the Fourth Military Medical University, Xian, Shanxi
  - Sichuan University West China Hospitcal, Chengdu, Sichuan
  - Peking University People's Hospital, Beijing
  - PekingTongren Hospital, Beijing
  - Eye & ENT Hospital of Fudan University, Shanghai
  - Shanghai First People's Hospital, Shanghai